CLINICAL TRIAL: NCT07209501
Title: Evaluating the Feasibility and Acceptability of Inhalation Aromatherapy for Reducing Chemotherapy-Induced Nausea and Vomiting (CINV) in Patients Undergoing Autologous Haematopoietic Stem Cell Transplant (HSCT): A Pilot Study
Brief Title: Evaluating the Feasibility and Acceptability of Inhalation Aromatherapy for Patients Undergoing Autologous Haematopoietic Stem Cell Transplant (HSCT)
Acronym: Aroma-CINV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-3551; 2024AMII-Aug03 (Other Grant/Funding Number: SINGHEALTH DUKE-NUS ACADEMIC MEDICINE INNOVATION INSTITUTE (AMII) NURSING INNOVATION GRANT 2024)
Record Dates: First submitted 2025-10-02; First posted 2025-10-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
Keywords: aromatherapy; Chemotherapy-Induced Nausea and Vomiting; Autologous Haematopoietic Stem Cell Transplant
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants in the control group will receive the placebo intervention in addition to standard care. Participants will be provided with an identical aromatherapy inhaler stick infused solely with jojoba oil. Jojoba oil, primarily used as a carrier oil for dilution, has little to- no scent and no known therapeutic or anxiolytic effects when inhaled. This ensures that any potential benefits observed in the intervention group can be attributed to the active essential oil blends rather than the inhalation process itself.
  Interventions: Other: Aromatherapy inhaler (placebo)
- Intervention group (Active Comparator): Participants in the intervention group will receive inhalation therapy via an aromatherapy inhaler stick*, on top of standard care.
  Participants will be instructed to use the inhaler stick every four hours when they are awake, and whenever they feel nauseous, by holding the inhaler stick a finger's length away from their nostrils and inhaling through one nostril at a time. Each administration should not last more than 5 minutes. Participants will commence using the inhaler stick on the day of chemotherapy, until five days after the completion of chemotherapy (a total of six days).
  Interventions: Other: Aromatherapy inhaler

INTERVENTIONS:
Other: Aromatherapy inhaler — Participants in the intervention group will receive inhalation therapy via an aromatherapy inhaler stick*, on top of standard care. Participants will be instructed to use the inhaler stick every four hours when they are awake, and whenever they feel nauseous, by holding the inhaler stick a finger's length away from their nostrils and inhaling through one nostril at a time. Each inhaler administration should not last more than 5 minutes. Participants will commence using the inhaler stick on the day of chemotherapy, until five days after the completion of chemotherapy (total of six days). Given the subjective nature of scents, participants in the intervention group will be given a choice between two therapeutic aroma blends - N1 and N2 - before commencing the study. This approach aims to minimize the risk of negative associations with a particular scent and enhance participant adherence to the intervention.
  Arms: Intervention group
Other: Aromatherapy inhaler (placebo) — Participants in the control group will receive the placebo intervention in addition to standard care. They will be provided with an identical aromatherapy inhaler stick infused solely with jojoba oil. Jojoba oil, primarily used as a carrier oil for dilution, has littleto- no scent and no known therapeutic or anxiolytic effects when inhaled.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate whether aromatherapy inhaler sticks can reduce nausea and vomiting in patients receiving chemotherapy as part of their stem cell transplant treatment. The main questions it aims to answer are:

* Can aromatherapy inhaler sticks be practically used by patients undergoing stem cell transplant (feasibility)?
* Do patients find aromatherapy inhaler sticks acceptable to use during their treatment?
* How effective are aromatherapy inhaler sticks at reducing chemotherapy-induced nausea and vomiting?
* What are patients' experiences when using aromatherapy during stem cell transplant?

Researchers will compare patients using aromatherapy inhaler sticks with essential oils to patients using inhaler sticks with only jojoba oil (placebo) to see if the essential oils provide additional benefits for reducing nausea and vomiting.

Participants will:

* Use their assigned inhaler stick every four hours when awake and whenever they feel nauseous
* Hold the inhaler stick a finger's length from their nostrils and inhale through one nostril at a time
* Use the inhaler stick for no more than 5 minutes per session
* Begin using the inhaler on the day of chemotherapy and continue until five days after chemotherapy completion (total of six days)
* Receive standard care for nausea and vomiting alongside the inhaler stick
* Complete study journals to record their experiences This is a single-blinded study, meaning participants will not know whether they received the aromatherapy or placebo inhaler stick.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years and older
* Able to provide informed consent
* Admitted for autologous stem cell transplant receiving melphalan conditioning chemotherapy regime
* Willing to have interviews audio-recorded

Exclusion Criteria:

* Currently using essential oils of any form (e.g. diffuser, topical application,
* Known sensitivity/ allergy to essential oils
* Any olfactory impairments (i.e. conditions that impair or alter sense of smell - for example, allergic rhinitis, chronic lung disease, blocked nose)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From commencement of study (Day 1) to the end of treatment (Day 6)
  Percentage of eligible patients who consent to join the study will be measured to evaluate the feasibility of using inhalation aromatherapy to reduce chemotherapy-induced nausea and vomiting (CINV) for patients undergoing haematopoietic stem cell transplant (HSCT)
Retention Rate | From commencement of study (Day 1) to the end of treatment (Day 6)
  Percentage of participants who complete the study will be measured to evaluate the feasibility of using inhalation aromatherapy to reduce chemotherapy-induced nausea and vomiting (CINV) for patients undergoing haematopoietic stem cell transplant (HSCT)
Adherence rate | From commencement of study (Day 1) to the end of treatment (Day 6)
  Percentage of participants in the intervention group who use the inhaler stick as instructed measured to evaluate the feasibility of using inhalation aromatherapy to reduce chemotherapy-induced nausea and vomiting (CINV) for patients undergoing haematopoietic stem cell transplant (HSCT)
Patient-reported satisfaction | From commencement of study (Day 1) to the end of treatment (Day 6)
  Measured through Likert-scale items at the end of the study to evaluate the acceptability of using inhalation aromatherapy to reduce chemotherapy-induced nausea and vomiting (CINV) for patients undergoing hematopoietic stem cell transplant (HSCT). The Feasibility of intervention Likert-scale and the Acceptability of intervention Liker-scale will be used. The Likert-scale consist of a rating of 1- 5 where 1 is strongly disagree and 5 is strongly agree and to be rated by participants.
Perceptions and Overall Experience | From commencement of study (Day 1) to the end of treatment (Day 6)
  Qualitative insights from semi-structured interviews on ease of use, perceived helpfulness and overall experience to evaluate acceptability of using inhalation aromatherapy to reduce chemotherapy-induced nausea and vomiting (CINV) for patients undergoing haematopoietic stem cell transplant (HSCT)

SECONDARY OUTCOMES:
Severity of Nausea | From commencement of study (Day 1) to the end of treatment (Day 6)
  Patient-reported nausea severity measured daily using a Visual Analog Scale (VAS, 0 = no nausea, 10 = worst possible nausea).
Frequency of Vomiting | From commencement of study (Day 1) to the end of treatment (Day 6)
  Number of vomiting episodes recorded in patient journals and verified against electronic medical records
Use of Rescue Anti-Emetics | From commencement of study (Day 1) to the end of treatment (Day 6)
  Frequency and dosage of rescue anti-emetic medication administered, retrieved from electronic medical records
Oral Intake | From commencement of study (Day 1) to end of treatment (Day 6)
  Daily oral intake as documented in medical records as an indicator of nausea levels
Grading of Chemotherapy-Induced Nausea and Vomiting (CINV) | From commencement of study (Day 1) to end of treatment (Day 6)
  Grading of CINV severity using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) on a 0-4 scale, where higher scores indicate more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Tay, Bachelor of Nursing, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided